CLINICAL TRIAL: NCT01355575
Title: RiFL: Rifaximin in Fatty Liver Disease. Does Modulation of Gut Microbiota Reduce Hepatic Inflammation in Non-Alcoholic Steatohepatitis (NASH)?
Brief Title: Rifaximin in Fatty Liver Disease
Acronym: RiFL
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Primary endpoint data review concluded no further patients required.
Sponsor: Imperial College London (Other)
Collaborators: National Health Service, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-021515-17; 2010-021515-17 (EudraCT Number); 10/H0711/58 (Other: Research Ethics Committee); 45706 (Other: Imperial Joint Research Office)
Record Dates: First submitted 2011-05-17; First posted 2011-05-18 (Estimated); Results first posted 2020-09-04 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Nonalcoholic Fatty Liver Disease; NAFLD; Nonalcoholic Steatohepatitis
Keywords: Microbiota; Insulin resistance; Bacterial endotoxin; Hepatic triglyceride; Inflammation
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Insulin Resistance; Inflammation | interventions — Rifaximin

STUDY DESIGN:
Intervention Model Description: An open label pilot study with two phases (rather than 2 arms). All patients receiving 6 weeks Rifaximin 400mg twice daily, followed by a 6 week observation period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rifaximin for 6-weeks followed by 6-week observation period (Experimental): All patients receiving 6 weeks Rifaximin 400mg twice daily, followed by a 6 week observation period.
  Interventions: Drug: Rifaximin

INTERVENTIONS:
Drug: Rifaximin — Rifaximin tablet, oral administration, 400mg twice daily for 6 weeks.
  Other Names: Xifaxan

SUMMARY:
TITLE Rifaximin in Fatty Liver Disease (RiFL) DESIGN Open-label pilot study HYPOTHESIS Reduction in gut flora by the antibiotic Rifaximin reduces hepatic inflammation in Non-Alcoholic Steatohepatitis (NASH).

AIMS To provide proof-of-concept data on the therapeutic potential of gut flora modification in NASH OUTCOME MEASURES

Primary:

• Change in serum ALT from baseline by 25 IU/L or to within normal range after 6 weeks of Rifaximin therapy

Secondary:

* Change in intrahepatic triglyceride, estimated by in vivo proton magnetic resonance spectroscopy (1H MRS)
* Change in hepatic insulin resistance, estimated by the hyperinsulinaemic euglycaemic clamp
* Changes to the faecal bacterial microbiome assessed by faecal DNA pyrosequencing and fluorescent in-situ hybridisation (FISH)
* Differences in urinary metabolic profiles as assessed by high-resolution proton nuclear magnetic resonance spectroscopy

POPULATION Patients with biopsy-confirmed non-alcoholic steatohepatitis and persistently raised serum aminotransferase levels

TREATMENT The non-absorbable antibiotic Rifaximin DURATION This was an open-label study of Rifaximin (Normix, Alfa Wasserman S.p.A, Bologna, Italy) 400mg twice daily for six weeks followed by a further six weeks observation period during which patients received standard care.

DETAILED DESCRIPTION:
STUDY OBJECTIVES The primary endpoint was change in ALT after 6 weeks of Rifaximin. Secondary endpoints were change in hepatic lipid content and insulin sensitivity measured with a hyperinsulinaemic euglycaemic clamp.

STUDY DESIGN This was an open-label study of Rifaximin (Normix, Alfa Wasserman S.p.A, Bologna, Italy) 400mg twice daily for six weeks followed by a further six weeks observation period during which patients received standard care. Compliance with treatment was checked by collection of empty blister packs. Subjects were asked to provide a structured dietary and lifestyle history as previously described (Williams HR, Cox IJ, Walker DG, North BV, Patel VM, Marshall SE, Jewell DP, et al. Characterization of inflammatory bowel disease with urinary metabolic profiling. Am J Gastroenterol 2009;104:1435-1444). The primary endpoint was change in ALT after 6 weeks' Rifaximin therapy. Secondary endpoints were change in hepatic and whole-body insulin sensitivity assessed by the two-stage hyperinsulinaemic euglycaemic clamp and change in hepatic triglyceride content assessed by proton nuclear magnetic resonance spectroscopy at 6 weeks from baseline. Serum ALT, biochemistry and anthropometrics were also measured at 12 weeks to look for longer-term effects. Stool microbiota, urinary metabolic profile and serum cytokine profile were measured before and after intervention.

PARTICIPANT ENTRY

INCLUSION CRITERIA Male and female patients were eligible for inclusion if aged between 18 and 70 years with non-alcoholic steatohepatitis histologically-proven, as evidenced by the presence of all of: steatosis, hepatocyte ballooning and lobular inflammation, and scored according to Kleiner(18) by a single experienced histopathologist (RDG) within the previous year, with or without mild to moderate fibrosis (stage 0-3/4) and with persistently elevated alanine aminotransferase (ALT) values on at least two occasions in the three months prior to recruitment.

EXCLUSION CRITERIA Patients were excluded if there was histological evidence of cirrhosis; hepatic decompensation; regular alcohol consumption exceeding 14 units/week (16g ethanol/day) for a woman or 21 units/week (24g ethanol/day) for a man; evidence of viral, autoimmune or other metabolic liver disease on a chronic liver disease screen; a history of malignancy or systemic inflammatory conditions; myocardial infarction or cerebrovascular events in the preceding 6 months; a history of bariatric surgery, blind loop or short bowel; use of any treatment known or suspected to change bowel flora within 3 months of enrolment; initiation or major dose change of metformin, thiazolinediones, biguanides, statins, fibrates, anti-obesity medications or insulin within 3 months of enrolment.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided written informed consent prior to screening
* Men and women aged 18-70 years
* With non-alcoholic steatohepatitis histologically-proven, as evidenced by the presence of all of: steatosis, hepatocyte ballooning and lobular inflammation, and scored according to Kleiner(18) by a single experienced histopathologist (RDG) within the previous year, with or without mild to moderate fibrosis (stage 0-3/4)
* With persistently elevated alanine aminotransferase (ALT) values on at least two occasions in the three months prior to recruitment

Exclusion Criteria:

* NAFLD with cirrhosis (fibrosis score 4)
* Other causes of chronic liver disease

  * Viral hepatitis (HBV, HCV negative)
  * Alcohol intake >14units/week (women) or >21units/week (men)
  * Haemachromatosis (abnormal transferrin saturation, haemochromatosis genotyping)
* Evidence of hepatic decompensation

  * Ascites
  * Hepatic encephalopathy
  * Abnormal total bilirubin (except patients with Gilbert's syndrome), albumin, prolonged prothrombin time, low platelets)
  * Oesophageal or gastric varices
* Moderate or severe renal dysfunction (CKD3+, estimated GFR <60ml/min/1.73m2)
* Hepatocellular carcinoma
* Primary metabolic causes of hepatic steatosis (e.g. familial hypertriglyceridaemia, abetalipoproteinaemia)
* Other malignancy
* Pregnant or lactating women or women of childbearing potential unwilling/unable to use adequate contraceptive methods
* Systemic inflammatory conditions

  * Arthritis
  * Connective tissue disorders
  * Inflammatory bowel disease
* Myocardial infarction within 6 months
* Stroke within 6 months
* Bariatric surgery/ blind loop/ short bowel
* Treatment known/suspected to change gut flora (e.g. systemic antibiotics, colestyramine, lactulose, polyethylene glycol) within 3 months
* Treatment with drugs known to cause hepatic steatosis (e.g. corticosteroids, HAART, amiodarone, high dose oestrogens, tamoxifen) within 3 months
* Initiation or major dose change of metformin, thiazolidinediones, biguanides, statins, fibrates, anti-obesity medications or insulin within 3 months of enrolment
* Patients with allergy to Rifaximin or Rifamycin
* Patients with a cardiac pacemaker, history of penetrating eye injury, metal foreign body or any other contra-indication to MRI scanning, as specified in the local MRI safety checklist
* Any other clinical, social or psychological issues which, in the opinion of the investigators may preclude satisfactory completion of the study protocol

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2011-05; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy FL Cobbold, PhD, Principal Investigator — Imperial College London; Mark R Thursz, MD, Study Chair — Imperial College London
Locations (1):
- Liver Unit, St Mary's Hospital, Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Rifaximin for 6-weeks Then Standard Care: Rifaximin for 6 weeks in addition to standard care, followed by 6 weeks observation period during which patients receive standard care.
  Rifaximin: Rifaximin tablet, oral administration, 400mg twice daily for 6 weeks.
Period: Overall Study
Arm/Group | Rifaximin for 6-weeks Then Standard Care
Started | 15
Completed | 13
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Groups:
- Patients Combined: All patients in one group
Arm/Group | Patients Combined
Number analyzed (Participants) | 15
Age, Continuous [Median (Full Range); unit: years] | 46 [32 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 13

OUTCOME MEASURES:

1. Primary Outcome: Serum Alanine Aminotransferase (ALT) Levels
Description: Alanine aminotransferase (ALT) after 6-weeks of Rifaximin from baseline (end of treatment) and 12 weeks (6 weeks after end of treatment).
  ALT values reported are the values from 6-weeks Rifaximin treatment compared to baseline, and ALT values from 12 weeks (after 6 weeks of SoC) compared to baseline.
Time Frame: Baseline, 6 weeks (end of treatment) and 12 weeks (6 weeks after end of treatment)
Measure: Median (Full Range); unit: iu/L
Groups:
- Rifaximin for 6-weeks: Phase 1 Rifaximin: Rifaximin tablet, oral administration, 400mg twice daily for 6 weeks.
- Standard of Care for 6-weeks: Phase 2 The 6-weeks Rifaximin treatment was followed by an observation period for 6-weeks during which patients received standard of care. All patients who had received Rifaximin for 6-weeks then received standard of care for the 6-week period.
Arm/Group | Rifaximin for 6-weeks | Standard of Care for 6-weeks
Number analyzed (Participants) | 15 | 15
iu/L | 63 [41 to 218] | 83 [30 to 217]

2. Secondary Outcome: Insulin Resistance
Description: Hepatic and systemic insulin resistance assessed using the hyperinsulinaemic euglycaemic clamp method.
  Measured in % Suppression of Endogenous Glucose Production (SEGP). Values reported are the value from baseline and value from 6 weeks Rifaximin treatment.
Time Frame: Baseline and 6 weeks (end of treatment)
Population: Data not collected during standard of care.
Measure: Median (Full Range); unit: % SEGP
Groups:
- Rifaximin Baseline: Rifaximin baseline
- Rifaximin After 6-weeks: Rifaximin: Patients received Rifaximin tablet, oral administration, 400mg twice daily for 6 weeks.
Arm/Group | Rifaximin Baseline | Rifaximin After 6-weeks
Number analyzed (Participants) | 14 | 14
% SEGP | 35.2 [15.3 to 51.7] | 30 [10.8 to 50.5]

3. Secondary Outcome: Hepatic Triglyceride Content
Description: In vivo proton magnetic resonance spectroscopy (1H MRS) to derive a T2-corrected triglyceride to water ratio (hepatic lipid content- intra-hepatocellular lipid (IHCL)).
  The values reported are the values from baseline and the values from 6 weeks Rifaximin treatment.
Time Frame: Baseline and 6 weeks (end of treatment)
Population: Data not collected during standard of care.
Measure: Median (Full Range); unit: % hepatic lipid content
Arm/Group | Rifaximin Baseline | Rifaximin After 6-weeks
Number analyzed (Participants) | 14 | 14
% hepatic lipid content | 21.6 [2.2 to 46.2] | 24.8 [1.7 to 59.3]

ADVERSE EVENTS:
Time Frame: 12 weeks
Groups:
- Rifaximin for 6-weeks: Participants received rifaximin tablet, oral administration, 400mg twice daily for 6-weeks.
- Standard of Care for 6-weeks: The 6-weeks Rifaximin treatment was followed by an observation period for 6-weeks during which patients received standard of care. All patients who had received Rifaximin for 6-weeks then received standard of care for the 6-week period.
Arm/Group | Rifaximin for 6-weeks | Standard of Care for 6-weeks
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 1/15 | 0/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rifaximin for 6-weeks (N=15) | Standard of Care for 6-weeks (N=15)
Loose stool (Gastrointestinal disorders) | 1 (1) | 0 (0) — 36 hours loose stool which resolved spontaneously and therapy was not discontinued.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes